CLINICAL TRIAL: NCT02997371
Title: A Randomised Double Blind Placebo Controlled Dose-range Study Using Placebo, 1.5g and 3.0g of Intravenous Recombinant Interleukin-1 Receptor Antagonist (Anakinra) for Patients With Moderate-to-severe TBI
Brief Title: IL-1ra Dose-range Study for Moderate-to-severe TBI Patients
Acronym: IL1ra
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adel Helmy (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Adel Helmy, MA, MB BChir, PhD, FRCS (SN), University of Cambridge
Organization: University of Cambridge (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCTU0185
Record Dates: First submitted 2016-12-07; First posted 2016-12-20 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Traumatic Brain INjury
Keywords: Traumatic brain injury; Microdialysis; Interleukin-1 receptor antagonist; Magnetic Resonance Imaging; Positron Emission Tomography
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Interleukin 1 Receptor Antagonist Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Isotonic saline administered as an injection and infusion
  Interventions: Drug: Isotonic saline
- 1.5 g Kineret (Experimental): Kineret provided as a 500 mg injection followed by a 1g infusion.
  Interventions: Drug: Anakinra Prefilled Syringe
- 3.0 g Kineret (Experimental): Kineret provided as a 500 mg injection followed by a 2.5g infusion.
  Interventions: Drug: Anakinra Prefilled Syringe

INTERVENTIONS:
Drug: Anakinra Prefilled Syringe — Administration as initially intravenous injection followed by a intravenous infusion
  Other Names: Kineret
  Arms: 1.5 g Kineret; 3.0 g Kineret
Drug: Isotonic saline — Placebo, administration as initially intravenous injection followed by a intravenous infusion
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Traumatic brain injury (TBI) is a common condition with high degree of morbidity and mortality (Hyder et al., 2007). Current treatment paradigms for TBI focus on mitigating secondary injury and maintaining cerebral physiology (Carney et al., 2016), however, there are currently no approved drugs that target the underlying conditions for patients suffering from TBI (Bullock et al., 1999). It is increasingly recognised that the innate inflammatory response to TBI may inflict injury (Lucas et al., 2006), and one of the most prominent mediators of inflammation in the injured brain is the Interleukin-1 (IL-1) receptor pathway (Allan et al., 2005). An endogenous antagonist to IL-1, is available in recombinant form (IL-1ra, Kineret), and is known to be safe in TBI (Helmy et al., 2014).

In order to fully understand, and potentially optimize, the effect of Kineret, the investigators wish to conduct a dose-response study by giving three cohorts (n=20 per group) either placebo (isotonic saline), 1.5g or 3.0g of active substance administered intravenously in a double-blind, randomized setting. The concentrations have in previous studies not been shown to present any side-effects (Singh et al., 2014). The drug will be provided within 12 hours after trauma. The goal will be to provide a dose-response effect on the cerebral inflammatory response. As secondary goals, the investigators will assess the brain damage by measuring proteins in blood and cerebrospinal fluid, functional outcome and inflammation in the brain using positron emission tomography.

DETAILED DESCRIPTION:
Aim

The hypothesis is that an increasing dose of the anti-inflammatory drug recombinant human Interleukin-1 receptor antagonist (IL-1ra, Kineret) will modulate the inflammatory state of the traumatically injured brain, which will attenuate the injurious processes that occur following TBI.

Study Design

While different doses of Anakinra have been used in trials, there is no knowledge of what constitutes an optimized concentration of the drug. To address this limitation, the current study will be a dose-response study in a double blind randomised clinical fashion, using placebo (n=20), 1.5 g ("intermediate dose") or (n=20) and 3.0 g ("high dose")(n=20) of Anakinra provided the first 48 hours (drug/placebo administered initially as 500 mg infusion bolus and later as an 1g or 2.5g infusion for 48 hours). Thus, a total of n=60 patients will be included. Sample-size analyses have indicated that the number of patients is sufficient to detect differences in the inflammatory response as gauged with cytokine measurements using cerebral microdialysis.

As surrogate markers of outcome for these patients, several protein biomarkers of brain injury and proteins of the innate immune responses will be quantified using techniques called ELISA and multiplex assay technology. The investigators also wish to use radiological techniques, such as magnetic resonance imaging to study damages in white matter tracts in the brain and positron emission tomography to assess the degree of microglial activation. All these methods will be used to assess the potential benefit of the treatment vs placebo.

By this type of study design, it will minimize bias and confounders that may influence the study.

Patient Recruitment

Patients with a clinical diagnosis of severe and moderate TBI will be identified by the research team at the daily departmental neuro-critical care unit meeting. Patients meeting the inclusion criteria will be approached for consent/assent if conscious or if next of kin is present. If not, consent will be assumed as we know Anakinra to be safe and there is likely to be a narrow therapeutic window. With the current patient load at Addenbrooke's Hospital, Cambridge, the investigators deem it possible to recruit one patient per week, thus estimating that the recruiting phase will take approximately two years to complete.

Sampling

All the sampling will be conducted during the acute phase when the patient is unconscious in the neuro-critical care unit. Microdialysis probes are sampled hourly. To assess inflammatory activity in the brain, positron emission tomography will be performed within the first week and after 2-3 weeks. Magnetic resonance imaging will be performed the first 2-3 weeks and then after 6 months. To measure the patient's adaptive immune response to brain specific proteins, specialised auto-immunisation assays will be performed on patient blood at day 1-3 following injury as well as after 2-3 weeks.

During the intensive care phase, blood and cerebrospinal fluid will be sampled twice per day (approximately 3mL per sampling time per compartment, volumes that we do not deem harmful to the patient) and will be collected together with hourly microdialysate fluid samples the first 7 days from admission. Blood will also be sampled at an outpatient clinic follow up at 6 and 12 months following injury. Patient samples will be anonymised and stored at -80degC in the Division of Neurosurgery, Department of Clinical Neurosciences, University of Cambridge before analysis.

It will not to be possible to measure cytokines, the drug and biomarkers from all microdialysis samples due to volume constraints. Moreover, we believe that a temporal resolution of 6 hours is probably adequate for the brain concentration of the drug while 12 hours is sufficient in serum. APP and tau will also be measured every 6 hours. The only parameter that will be hourly analysed in microdialysis is cytokine and chemokines through a luminex panel.

Clinical Follow-up

Patients will be followed up at a clinic visit at 6 and 12 months after trauma by questionnaire survey using standardised outcome measures in neurosurgical patients including the golden standard extended Glasgow Outcome Score and Short Form 36.

ELIGIBILITY:
Inclusion Criteria:

1. Suffer from a TBI, present with a Glasgow Coma Scale (GCS) of 3-13 and be deemed to be in need of neuro-critical care and intracranial monitoring for at least 72 hours.
2. Be aged 18-65
3. The first dose of Kineret (or placebo) must be provided within 12 hours after trauma.

Exclusion Criteria:

1. Head injury unlikely to survive 5 days (radiological evidence of above as judged by clinical team, bilateral fixed and dilated pupils).
2. Follow up not possible
3. Not suitable for insertion of cranial access device to monitor the brain (such as bleeding complications)
4. Active immunosuppression therapy (evidence of neutropenia, immunosuppression secondary to immunomodulatory medications, chemotherapy or radiation therapy in the 3 months preceding study entry)
5. Severe Renal Insufficiency or End Stage Renal Disease (defined as a creatinine clearance <30 ml/min)
6. Pregnancy/Nursing mothers
7. Known hypersensitivity to E. coli derived products
8. Administration of live vaccine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Decrease of pro-inflammatory cytokines in brain extracellular fluid (ECF) | First 48 hours
  Decrease of Tumor necrosis factor alpha and interferon gamma cytokines in brain ECF

SECONDARY OUTCOMES:
Patient outcome GOSe | 6 months and 12 months
  Extended Glasgow Outcome Score (GOSe) assessments at 6 months and 1 year.
Patient outcome SF36 | 6 months and 12 months
  Short Form - 36 (SF-36) assessments at 6 months and 1 year.
Imaging outcome - PET-MRI | During the first 14 days
  To determine degree of microglial activation globally and in the locality of the microdialysis catheter, using magnetic resonance imaging (MRI) in combination with positron emission tomography (PET) PK-11195 (an an isoquinoline carboxamide) ligand.
Imaging outcome - DTI-MRI | During the first 14 days
  To determine degree of axonal injury globally and in the locality of the microdialysis catheter, using magnetic resonance imaging (MRI) in combination with diffuse tensor imaging (DTI).
Biochemical outcome - S100B | During the first 7 days + at 6 months and 12 months
  Concentrations of protein biomarkers of tissue fate, S100B in serum (µg/L) twice per day as well as after 6 months and 12 months.
Biochemical outcome - NF-L | During the first 7 days
  Concentrations of protein biomarkers of tissue fate, Concentrations of protein biomarkers of tissue fate, Neurofilament Light (NF-L) in serum (µg/L) twice per day as well as after 6 months and 12 months.
Biochemical outcome - Tau | During the first 7 days
  Concentrations of protein biomarkers of tissue fate, microtubuli associated protein tau (tau) measured in microdialysis every 6 hours.
Biochemical outcome - APP | During the first 7 days
  Concentrations of protein biomarkers of tissue fate, Amyloid Precursor Protein Beta (APP) associated protein tau measured in microdialysis every 6 hours.
Biochemical outcome - Autoreactivity versus MBP | During the first 7 days + at 6 months and 12 months
  Concentration of circulating T-cells with autoreactivity towards myelin basic protein (MBP) in serum.
Monitoring outcome - ICP | First 7 days
  Intracranial pressure (ICP, mmHg) during the neuro-critical care unit (NCCU) stay.
Monitoring outcome - CPP | First 7 days
  Cerebral perfusion pressure (CPP, mmHg) during the NCCU stay.
Monitoring outcome - Cerebral Metabolism LPR | First 7 days
  Cerebral metabolism, by measuring lactate:pyruvate ratio (LPR) in microdialysis.
Monitoring outcome - Brain tissue oxygenation | First 7 days
  Brain tissue oxygen (mmHg).
Monitoring outcome - PRx | First 7 days
  Derived variables of cerebral elastance (Pressure reactivity index, PRx).
Pharmacological outcome - Concentration of IL1ra in brain tissue | First week
  IL-1ra brain concentration (pg/ml), measured every 6 hours by cerebral microdialysis.
Pharmacological outcome - Concentration of IL1ra in serum | First week
  IL-1ra serum concentration (pg/ml), measured every 12 hours.
Side effects of the IL1ra | First week + up to 12 months follow-up
  To study any potential side-effect of the drug, both known and unknown.

CONTACTS AND LOCATIONS:
Overall Officials: Adel Helmy, MA, MB BChir, FRCS, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospital NHS Trust, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Allan SM, Tyrrell PJ, Rothwell NJ. Interleukin-1 and neuronal injury. Nat Rev Immunol. 2005 Aug;5(8):629-40. doi: 10.1038/nri1664. PMID 16034365
- [Background] Bullock MR, Lyeth BG, Muizelaar JP. Current status of neuroprotection trials for traumatic brain injury: lessons from animal models and clinical studies. Neurosurgery. 1999 Aug;45(2):207-17; discussion 217-20. doi: 10.1097/00006123-199908000-00001. PMID 10449064
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000
- [Background] Helmy A, Guilfoyle MR, Carpenter KL, Pickard JD, Menon DK, Hutchinson PJ. Recombinant human interleukin-1 receptor antagonist in severe traumatic brain injury: a phase II randomized control trial. J Cereb Blood Flow Metab. 2014 May;34(5):845-51. doi: 10.1038/jcbfm.2014.23. Epub 2014 Feb 26. PMID 24569690
- [Background] Hyder AA, Wunderlich CA, Puvanachandra P, Gururaj G, Kobusingye OC. The impact of traumatic brain injuries: a global perspective. NeuroRehabilitation. 2007;22(5):341-53. PMID 18162698
- [Background] Lucas SM, Rothwell NJ, Gibson RM. The role of inflammation in CNS injury and disease. Br J Pharmacol. 2006 Jan;147 Suppl 1(Suppl 1):S232-40. doi: 10.1038/sj.bjp.0706400. PMID 16402109
- [Background] Singh N, Hopkins SJ, Hulme S, Galea JP, Hoadley M, Vail A, Hutchinson PJ, Grainger S, Rothwell NJ, King AT, Tyrrell PJ. The effect of intravenous interleukin-1 receptor antagonist on inflammatory mediators in cerebrospinal fluid after subarachnoid haemorrhage: a phase II randomised controlled trial. J Neuroinflammation. 2014 Jan 3;11:1. doi: 10.1186/1742-2094-11-1. PMID 24383930